CLINICAL TRIAL: NCT06870071
Title: Effect of Quadro-Iliac Plane Block on Quality of Recovery After Total Hip Arthroplasty: A Prospective, Randomized, Controlled, Double-Blind, Multicenter Study
Brief Title: Effect of Quadro-Iliac Plane Block on Recovery After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, M.D., Department of members Anesthesiology and Reanimation, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Quadro-Iliac Block Hip
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): IV paracetamol (1 g, 3×1) and IV dexketoprofen (50 mg, 2×1)
  Interventions: Other: Quadro iliac plane block
- Quadro iliac plane block (Active Comparator): 40 mL of 0.25% bupivacaine
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — IV paracetamol (1 g, 3×1) and IV dexketoprofen (50 mg, 2×1)
  Arms: Quadro iliac plane block
Other: Quadro iliac plane block — 40 mL of 0.25% bupivacaine
  Arms: control group

SUMMARY:
Total hip arthroplasty is a widely performed surgical procedure in the elderly population, aiming to relieve hip joint pain and restore function. Total hip arthroplasty is among the most critical surgical procedures in terms of morbidity and mortality within this demographic. To mitigate opioid-related adverse effects in this patient group, novel analgesic methods are needed. Regional anesthesia techniques used for postoperative pain management include epidural analgesia, lumbar plexus block, fascia iliaca block, femoral and obturator nerve blocks, and sacral erector spinae plane block. However, these procedures may result in complications such as epidural hematoma, postoperative headache, prolonged motor block, and extended hospital stay.

DETAILED DESCRIPTION:
Total hip arthroplasty is a widely performed surgical procedure in the elderly population, aiming to relieve hip joint pain and restore function. Total hip arthroplasty is among the most critical surgical procedures in terms of morbidity and mortality within this demographic. To mitigate opioid-related adverse effects in this patient group, novel analgesic methods are needed. Regional anesthesia techniques used for postoperative pain management include epidural analgesia, lumbar plexus block, fascia iliaca block, femoral and obturator nerve blocks, and sacral erector spinae plane block. However, these procedures may result in complications such as epidural hematoma, postoperative headache, prolonged motor block, and extended hospital stay.

Recently, Tulgar et al. introduced a novel fascial plane block called the "quadro-iliac plane block". This block is performed in the quadro-iliac plane, located between the inner surface of the iliac crest and the posterior surface of the quadratus lumborum muscle. In their study, Tulgar et al. bilaterally injected 40 mL of methylene blue into the quadro-iliac plane, observing widespread dye distribution along the posterior and anterior surfaces of the quadratus lumborum muscle, transversalis fascia, ilioinguinal, iliohypogastric, subcostal, and genitofemoral nerves, as well as the lumbar plexus. Based on these findings, quadro-iliac plane block has been proposed as a potentially effective technique for managing acute or chronic pain in the lumbosacral, abdominal, and hip regions. However, apart from a few case reports involving lumbar spine surgery and kidney transplantation, evidence regarding the efficacy of quadro-iliac plane block remains limited.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral THA.
* Spinal anesthesia.
* Age 18-85 years.
* ASA classification I-IV.

Exclusion Criteria:

* Patients who declined consent.
* Contraindications to regional anesthesia.
* Coagulation disorders.
* Infections at the block site.
* Emergency surgeries.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Postoperative Quality of Recovery-15 | 24 hours
  The primary outcome was the Quality of Recovery-15 score at 24 hours postoperatively. QoR-15 scores range from 0 to 150, with higher scores indicating better recovery quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)